CLINICAL TRIAL: NCT03434353
Title: A Phase 2, Randomized, Open-Label, Active-Controlled Study to Evaluate the Safety and Antiviral Activity of GS-9992 Plus Tenofovir Alafenamide (TAF) for 12 Weeks in Chronic Hepatitis B (CHB) Subjects
Brief Title: Study to Evaluate the Safety and Antiviral Activity of Inarigivir Soproxil (Formerly: GS-9992) Plus Tenofovir Alafenamide (TAF) for 12 Weeks in Adults With Chronic Hepatitis B (CHB)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to sponsor's decision to not pursue further development of inarigivir soproxil in chronic hepatitis B.
Sponsor: Gilead Sciences (Industry)
Collaborators: F-star Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-464-4437
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1: Inarigivir Soproxil 50 mg + TAF (Experimental): Viremic participants will be administered inarigivir soproxil 50 mg (2 x 25 mg capsules) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed by TAF 25 mg tablet once daily orally with food for 36 weeks.
  Interventions: Drug: Inarigivir Soproxil; Drug: TAF
- Group 2: TAF (Experimental): Viremic participants will be administered TAF 25 mg tablet once daily orally with food for 48 weeks.
  Interventions: Drug: TAF
- Group 3: Inarigivir Soproxil 200 mg + TAF (Experimental): Viremic participants will be administered inarigivir soproxil 200 mg (2 x 100 mg tablets) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed by TAF 25 mg tablet once daily orally with food for 36 weeks
  Interventions: Drug: Inarigivir Soproxil; Drug: TAF
- Group 4: Inarigivir Soproxil 100 mg + commercially available NUCs (Experimental): Virally suppressed participants receiving commercially available nucleoside/nucleotide (NUC) will be administered inarigivir soproxil 100 mg tablet once daily orally 1 hour before or 1 hour after a meal for 12 weeks. Participants will continue commercially available NUCs for 48 weeks.
  Interventions: Drug: Inarigivir Soproxil
- Group 5: Inarigivir Soproxil 400 mg + TAF (Experimental): Viremic participants will be administered inarigivir soproxil 400 mg (2 x 200 mg tablets) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed TAF 25 mg tablet once daily orally with food for 36 weeks.
  Interventions: Drug: Inarigivir Soproxil; Drug: TAF

INTERVENTIONS:
Drug: Inarigivir Soproxil — Administered orally once daily one hour before or one hour after a meal
  Other Names: SB 9200; GS-9992
  Arms: Group 1: Inarigivir Soproxil 50 mg + TAF; Group 3: Inarigivir Soproxil 200 mg + TAF; Group 4: Inarigivir Soproxil 100 mg + commercially available NUCs; Group 5: Inarigivir Soproxil 400 mg + TAF
Drug: TAF — Administered orally once daily with food
  Other Names: GS-7340; Vemlidy®
  Arms: Group 1: Inarigivir Soproxil 50 mg + TAF; Group 2: TAF; Group 3: Inarigivir Soproxil 200 mg + TAF; Group 5: Inarigivir Soproxil 400 mg + TAF

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of the 12 week treatment regimens of inarigivir soproxil plus tenofovir alafenamide (TAF) or commercially available nucleoside/nucleotide (NUC) in adults with chronic hepatitis B (CHB), to evaluate the antiviral activity of 12 weeks of inarigivir soproxil plus TAF versus TAF alone in viremic CHB participants (Groups 1-3, 5), and to evaluate the antiviral activity of 12 weeks of inarigivir soproxil with commercially available NUC(s) in virally suppressed CHB participants (Group 4).

ELIGIBILITY:
Key Inclusion Criteria:

* Groups 1-3 and 5:

  * Individuals not taking any prescribed hepatitis B virus (HBV) NUC treatment
* Group 4:

  * HBV deoxyribonucleic acid (DNA) ≤ 20 IU/mL at Screening by Central Lab.
  * Have been on a commercially available HBV NUC treatment(s)

Key Exclusion Criteria:

* Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus (HDV).
* Extensive bridging fibrosis or cirrhosis
* Evidence of hepatocellular carcinoma on imaging
* Any history of, or current evidence of, clinical hepatic decompensation (e.g., ascites, encephalopathy or variceal hemorrhage).
* Chronic liver disease of a non-HBV etiology
* Current alcohol or substance abuse

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince Margaret Hospital, Hong Kong
  - Prince of Wales Hospital-HK, Hong Kong
- South Korea (10):
  - Korea University Ansan Hospital, Ansan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Inje University Ilsan Paik Hospital, Ilsan
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Catholic University of Korea, Seoul Saint Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lim YS, Hui AJ, Jang JW, Tak WY, Ahn SH, Jang BK, et al. Safety, efficacy, & pharmacodynamic (PD) activity of 12 weeks treatment with oral RIG-I agonist, inarigivir (IRIG), plus 48 weeks of tenofovir alafenamide in adult patients with chronic hepatitis B: a phase 2 collaboration study [Abstract PO-2422]. The International Liver Congress: European Association for the Study of the Liver (EASL) Virtual; 2021 23-26 June.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Hong Kong and South Korea. The first participant was screened on 28 February 2018. The last study visit occurred on 26 January 2021.
Pre-assignment Details: 161 participants were screened.
Groups:
- Group 1: Inarigivir Soproxil 50 mg + TAF: Viremic participants were administered inarigivir soproxil 50 mg (2 x 25 mg capsules) once daily orally 1 hour before or 1 hour after a meal plus tenofovir alafenamide (TAF) 25 mg tablet once daily orally with food for 12 weeks followed by TAF 25 mg tablet once daily orally with food for 36 weeks.
- Group 2: TAF: Viremic participants were administered TAF 25 mg tablet once daily orally with food for 48 weeks.
- Group 3: Inarigivir Soproxil 200 mg + TAF: Viremic participants were administered inarigivir soproxil 200 mg (2 x 100 mg tablets) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed by TAF 25 mg tablet once daily orally with food for 36 weeks.
- Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s): Virally suppressed participants who were receiving commercially available nucleoside/nucleotide (NUC[s]) were administered inarigivir soproxil 100 mg tablet once daily orally 1 hour before or 1 hour after a meal for 12 weeks. Participants continued commercially available NUC(s) for 48 weeks.
- Group 5: Inarigivir Soproxil 400 mg + TAF: Viremic participants were administered inarigivir soproxil 400 mg (2 x 200 mg tablets) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed TAF 25 mg tablet once daily orally with food for 36 weeks.
Period: Overall Study
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s) | Group 5: Inarigivir Soproxil 400 mg + TAF
Started | 30 | 12 | 30 | 21 | 30
Completed | 16 | 9 | 16 | 18 | 12
Not Completed | 14 | 3 | 14 | 3 | 18
Not completed — Started commercial Hepatitis B virus therapy | 10 | 3 | 11 | 3 | 17
Not completed — Withdrew consent | 1 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Groups:
- Group 1: Inarigivir Soproxil 50 mg + TAF: Viremic participants were administered inarigivir soproxil 50 mg (2 x 25 mg capsules) once daily orally 1 hour before or 1 hour after a meal plus TAF 25 mg tablet once daily orally with food for 12 weeks followed by TAF 25 mg tablet once daily orally with food for 36 weeks.
- Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s): Virally suppressed participants who were receiving NUC(s) were administered inarigivir soproxil 100 mg tablet once daily orally 1 hour before or 1 hour after a meal for 12 weeks. Participants continued commercially available NUC(s) for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s) | Group 5: Inarigivir Soproxil 400 mg + TAF | Total
Number analyzed (Participants) | 30 | 12 | 30 | 21 | 30 | 123
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 23 | 5 | 19 | 11 | 13 | 71
  ≥50 years | 7 | 7 | 11 | 10 | 17 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 11 | 9 | 11 | 46
  Male | 18 | 9 | 19 | 12 | 19 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 12 | 30 | 21 | 30 | 123
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 30 | 12 | 30 | 21 | 30 | 123
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 8 | 5 | 22 | 11 | 30 | 76
  South Korea | 22 | 7 | 8 | 10 | 0 | 47
Hepatitis B Surface Antigen (HBsAg) Category [Count of Participants; unit: Participants]
  ≤ 4 log10 IU/mL | 16 | 4 | 23 | 19 | 21 | 83
  > 4 log10 IU/mL | 14 | 8 | 7 | 2 | 9 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 0.5 log10 IU/mL Decline in HBsAg From Baseline at Week 12 (Groups 1-3 and 5)
Time Frame: Baseline, Week 12
Population: The Full Analysis Set included all participants who were randomized to Groups 1 or 2, or enrolled in Group 3 and 5, and who took at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 30 | 12 | 30 | 30
percentage of participants | 23.3 [9.9 to 42.3] | 25.0 [5.5 to 57.2] | 0 [0.0 to 11.6] | 6.7 [0.8 to 22.1]
Statistical Analysis 1: Comparison: Group 1: Inarigivir Soproxil 50 mg + TAF vs Group 2: TAF; Test type: Other; Percentage Difference = -2.0, 95% CI 2-sided [-30.4 to 26.4] — The percentage difference (Group 1 - Group 2) & corresponding 2-sided 95% confidence interval (CI) were calculated by using stratum-adjusted Mantel-Haenszel proportions, stratified by baseline hepatitis B e antigen (HBeAg) status (positive,negative)
Statistical Analysis 2: Comparison: Group 2: TAF vs Group 3: Inarigivir Soproxil 200 mg + TAF; Test type: Other; Percentage Difference = -24.7, 95% CI 2-sided [-49.2 to -0.2] — The percentage difference (Group 3 - Group 2) and the corresponding 2-sided 95% CI were calculated by using stratum-adjusted Mantel-Haenszel proportions, stratified by baseline HBeAg status (positive, negative)
Statistical Analysis 3: Comparison: Group 2: TAF vs Group 5: Inarigivir Soproxil 400 mg + TAF; Test type: Other; Percentage Difference = -17.8, 95% CI 2-sided [-43.7 to 8.2] — The percentage difference (Group 5 - Group 2) and the corresponding 2-sided 95% CI were calculated by using stratum-adjusted Mantel-Haenszel proportions, stratified by baseline HBeAg status (positive, negative)

2. Primary Outcome: Percentage of Participants With ≥ 0.5 log10 IU/mL Decline in HBsAg From Baseline at Week 12 (Group 4)
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (Group 4) included all participants who were enrolled in Group 4, and who took at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s): Virally suppressed participants who were receiving commercially available NUC(s) were administered inarigivir soproxil 100 mg tablet once daily orally 1 hour before or 1 hour after a meal for 12 weeks. Participants continued commercially available NUC(s) for 48 weeks.
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 21
percentage of participants | 0 [0.0 to 16.1]

3. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in HBsAg From Baseline at Week 12 (Groups 1 Through 3 and 5)
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set (Group 1-3 and 5) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 30 | 12 | 30 | 30
percentage of participants | 0 [0.0 to 11.6] | 16.7 [2.1 to 48.4] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6]
Statistical Analysis 1: Comparison: Group 1: Inarigivir Soproxil 50 mg + TAF vs Group 2: TAF; Test type: Other; Percentage Difference = -16.6, 95% CI 2-sided [-37.7 to 4.4] — The percentage difference (Group 1 - Group 2) and the corresponding 2-sided 95% CI were calculated by using stratum-adjusted Mantel-Haenszel proportions, stratified by baseline HBeAg status (positive, negative)
Statistical Analysis 2: Comparison: Group 2: TAF vs Group 3: Inarigivir Soproxil 200 mg + TAF; Test type: Other; Percentage Difference = -16.9, 95% CI 2-sided [-38.1 to 4.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Group 2: TAF vs Group 5: Inarigivir Soproxil 400 mg + TAF; Test type: Other; Percentage Difference = -16.7, 95% CI 2-sided [-37.9 to 4.4] — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Percentage of Participants With ≥ 1 log10 IU/mL Decline in HBsAg From Baseline at Week 12 (Group 4)
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set (Group 4) were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 21
percentage of participants | 0 [0.0 to 16.1]

5. Secondary Outcome: Percentage of HBeAg-positive Participants Who Achieved HBeAg Loss and Seroconversion at Weeks 12, 24, 36, and 48 (Groups 1 Through 3 and 5)
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at post-baseline visit. HBeAg seroconversion was defined as HBeAb changing from negative or missing at baseline to positive at any postbaseline visit. Participants who had missing information were assumed to have no HBeAg loss and no HBeAg seroconversion.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Participants in the Full Analysis Set (Group 1-3 and 5) with HBeAg-positive status at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 18 | 7 | 14 | 16
percentage of participants
  Week 12 | 5.6 | 0 | 0 | 0
  Week 24 | 5.6 | 0 | 0 | 0
  Week 36 | 5.6 | 0 | 0 | 0
  Week 48 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of HBeAg-positive Participants Who Achieved HBeAg Loss and Seroconversion at Weeks 12, 24, 36, and 48 (Group 4)
Description: as for outcome 5
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Participants in the Full Analysis Set (Group 4) with HBeAg-positive status at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 7
percentage of participants
  Week 12 | 14.3
  Week 24 | 14.3
  Week 36 | 14.3
  Week 48 | 14.3

7. Secondary Outcome: Percentage of Participants Who Achieved HBsAg Loss at Weeks 12, 24, 36, and 48 (Groups 1 Through 3 and 5)
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at post-baseline visit. Participants who had missing information were assumed to have no HBeAg loss.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Participants in the Full Analysis Set (Groups 1 through 3 and 5) were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 30 | 12 | 30 | 30
percentage of participants
  Week 12 | 0 | 0 | 0 | 0
  Week 24 | 0 | 0 | 0 | 0
  Week 36 | 0 | 0 | 0 | 0
  Week 48 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Achieved HBsAg Loss at Weeks 12, 24, 36, and 48 (Group 4)
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at post-baseline visit.
Time Frame: Baseline, Weeks 12, 24, 36, and 48
Population: Participants in the Full Analysis Set (Group 4) were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 21
percentage of participants
  Week 12 | 0
  Week 24 | 0
  Week 36 | 0
  Week 48 | 0

9. Secondary Outcome: Number of Participants With Sequence Changes From Baseline Within the HBV Polymerase for Participants Who Had HBV DNA ≥ 69 IU/mL (Groups 1 Through 3 and 5)
Time Frame: Baseline, Week 48
Population: Participants with at least 12 weeks and 48 weeks of exposure to inarigivir soproxil and TAF, respectively, and with HBV DNA ≥ 69 IU/mL at Week 48 or Early Discontinuation were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 6 | 3 | 5 | 9
Participants | 4 | 0 | 0 | 4

10. Secondary Outcome: Percentage of Participants Experiencing Hepatitis B Virus (HBV) Virologic Breakthrough During 12 Weeks of Inarigivir Soproxil Treatment (Group 4)
Description: Virologic breakthrough was defined as HBV deoxyribonucleic acid (DNA) ≥69 IU/mL for 2 consecutive visits
Time Frame: Baseline up to Week 12
Population: Participants in the Full Analysis Set (Group 4) were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 21
percentage of participants | 0

11. Secondary Outcome: Change From Baseline in HBV DNA at Weeks 12, 16, 24, 36, and 48 (Groups 1 Through 3 and 5)
Time Frame: Baseline, Weeks 12, 16, 24, 36, and 48
Population: Participants in the Full Analysis Set (Groups 1-3 and 5) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 30 | 12 | 30 | 30
log10 IU/mL
  Baseline | 7.06 (1.530) | 7.06 (1.757) | 6.30 (1.365) | 6.61 (1.479)
  Change at Week 12: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 12 | -4.18 (0.959) | -4.24 (1.340) | -4.02 (0.854) | -3.93 (0.817)
  Change at Week 16: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 16 | -4.58 (1.023) | -4.65 (1.326) | -4.29 (0.946) | -4.23 (0.869)
  Change at Week 24: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 24 | -5.02 (1.101) | -5.25 (1.510) | -4.67 (1.049) | -4.76 (1.013)
  Change at Week 36: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 36 | -5.27 (1.194) | -5.53 (1.610) | -4.78 (1.207) | -4.92 (1.129)
  Change at Week 48: number analyzed (Participants) | 29 | 11 | 30 | 29
  Change at Week 48 | -5.36 (1.225) | -5.25 (1.839) | -4.83 (1.162) | -4.93 (1.370)

12. Secondary Outcome: Change From Baseline in HBsAg at Weeks 12, 16, 24, 36, and 48 (Groups 1 Through 3 and 5)
Time Frame: Baseline, Weeks 12, 16, 24, 36, and 48
Population: Participants in the Full Analysis Set (Groups 1-3 and 5) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 5: Inarigivir Soproxil 400 mg + TAF
Number analyzed (Participants) | 30 | 12 | 30 | 30
log10 IU/mL
  Baseline | 3.933 (0.8058) | 4.118 (0.6543) | 3.529 (0.8835) | 3.418 (0.8075)
  Change at Week 12: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 12 | -0.244 (0.3443) | -0.435 (0.5320) | 0.016 (0.2850) | -0.026 (0.3805)
  Change at Week 16: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 16 | -0.282 (0.3954) | -0.479 (0.5429) | 0.014 (0.2916) | -0.082 (0.4262)
  Change at Week 24: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 24 | -0.310 (0.4303) | -0.482 (0.5119) | -0.021 (0.3171) | -0.104 (0.5000)
  Change at Week 36: number analyzed (Participants) | 30 | 12 | 30 | 29
  Change at Week 36 | -0.330 (0.4363) | -0.524 (0.5430) | -0.055 (0.4213) | -0.209 (0.5319)
  Change at Week 48: number analyzed (Participants) | 29 | 11 | 30 | 29
  Change at Week 48 | -0.322 (0.4311) | -0.517 (0.5617) | -0.045 (0.4778) | -0.235 (0.5429)

13. Secondary Outcome: Change From Baseline in HBsAg at Weeks 12, 16, 24, 36, and 48 (Group 4)
Time Frame: Baseline, Weeks 12, 16, 24, 36, and 48
Population: Participants in the Full Analysis Set (Group 4) were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s)
Number analyzed (Participants) | 21
log10 IU/mL
  Baseline | 3.211 (0.5536)
  Change at Week 12 | -0.017 (0.0417)
  Change at Week 16 | -0.010 (0.0645)
  Change at Week 24 | -0.039 (0.0925)
  Change at Week 36 | -0.037 (0.0939)
  Change at Week 48 | -0.073 (0.1120)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization/enrollment up to Week 48 + 3 days Adverse events: Groups 1, 2, 3, 5: From first dose up to Week 48 + 3 days Group 4: From first dose up to Week 12 + 30 days (for Group 4, adverse events were planned to be collected only up to Week 12 + 30 days)
Description: All cause mortality: The All Randomized/Enrolled Analysis Set included all participants who were randomized (Group 1 and 2) or enrolled (Group 3-5) in the study.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Arm/Group | Group 1: Inarigivir Soproxil 50 mg + TAF | Group 2: TAF | Group 3: Inarigivir Soproxil 200 mg + TAF | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s) | Group 5: Inarigivir Soproxil 400 mg + TAF
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/12 | 0/30 | 0/21 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/12 | 1/30 | 0/21 | 1/30
Other Adverse Events (participants affected / at risk) | 8/30 | 7/12 | 15/30 | 9/21 | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Inarigivir Soproxil 50 mg + TAF (N=30) | Group 2: TAF (N=12) | Group 3: Inarigivir Soproxil 200 mg + TAF (N=30) | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s) (N=21) | Group 5: Inarigivir Soproxil 400 mg + TAF (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Inarigivir Soproxil 50 mg + TAF (N=30) | Group 2: TAF (N=12) | Group 3: Inarigivir Soproxil 200 mg + TAF (N=30) | Group 4: Inarigivir Soproxil 100 mg + Commercially Available NUC(s) (N=21) | Group 5: Inarigivir Soproxil 400 mg + TAF (N=30)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Influenza like illness (General disorders) | 0 | 0 | 2 | 6 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 6 | 1 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 3 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03434353/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT03434353/SAP_001.pdf